CLINICAL TRIAL: NCT02560610
Title: The Effect of OC000459 on Eosinophilic Airway Inflammation and Asthma Control in Subjects With Refractory Eosinophilic Asthma: a Randomised, Double-blind, Placebo Controlled Trial
Brief Title: Effect of OC000459 on Eosinophilic Airway Inflammation in Severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: Atopix Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OC000459/019/15; 2015-001833-26 (EudraCT Number)
Record Dates: First submitted 2015-09-04; First posted 2015-09-25 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Severe Eosinophilic Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia | interventions — (5-fluoro-2-methyl-3-quinolin-2-ylmethylindo-1-yl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OC000459 (Active Comparator): Once daily dose of 50mg OC000459 tablets orally for 12/24 weeks
  Interventions: Drug: OC000459
- Placebo (Placebo Comparator): Once daily dose of placebo tablets orally for 12/24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OC000459
  Arms: OC000459
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim is to study the effect of OC000459 on eosinophilic airway inflammation and asthma control in subjects with severe, refractory eosinophilic asthma.

DETAILED DESCRIPTION:
At week 12 subjects not on oral corticosteroids (OCS) will complete the treatment period and return after 4 weeks for final follow up visit. Those subjects who were taking OCS at baseline will continue for a maximum of 12 additional weeks, double blind period during which their current OCS treatment will be titrated down according to their clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Show evidence of reversible airflow obstruction documented within the previous 12 months or prior to Randomisation.
* Meet the European Respiratory Society/American Thoracic Society (ERS/ATS) criteria for severe asthma at Screening.
* Have documented evidence of eosinophilic airway inflammation during the 12 months prior to Screening.
* Have evidence of eosinophilic airway inflammation at Screening as reflected by an induced sputum eosinophil count of ≥3%.
* Subjects who are taking oral corticosteroids (OCS) must be receiving a 20 mg prednisolone equivalent dose, or less, daily for at least four weeks before the first dose of study drug. The dose of OCS should be unchanged for at least 14 days prior to the Baseline visit.

Exclusion Criteria:

* Treatment with XolairTM or anti-Th2 biologicals within 6 months prior to screening.
* Subjects with clinically significant abnormal serum biochemistry, haematology and urine examination values
* Subjects who have been hospitalised in the last 3 months.
* History of more than 2 episodes of confirmed bacterial lower respiratory tract infection or current lower respiratory tract infection.
* Subjects are current smokers or have a smoking history of >15 pack years.
* Significant comorbidity that in the Investigator's opinion is likely to impact the subject's participation in a 26 week study.
* Presence of a clinically important lung condition other than asthma, malignancy or previous history of cancer in remission for less than 12 months, clinically important liver or kidney disease, uncontrolled clinically significant cardiovascular disease, hypereosinophilic syndromes such as Churg-Strauss Syndrome or eosinophilic oesophagitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Compare the effect of OC000459 50mg given once daily with placebo on the induced sputum eosinophil counts. | Mean change from baseline and week 12

SECONDARY OUTCOMES:
The effect on pre- and post-bronchodilator spirometry using forced expiratory volume in one second (FEV1). | Every 4 weeks up to week 12
The effect of OC000459 on fractional exhaled nitric oxide (FeNO). | At 4,8 and 12 weeks
Measuring quality of life using standardised asthma quality of life questionnaire (AQLQ(S)). | At weeks 4,8 and 12
Statistical comparison from baseline on induced sputum eosinophil count. | At weeks 4,8 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Ian Pavord, Professor, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2015-001833-26/results